CLINICAL TRIAL: NCT03227900
Title: The Effect of lidocaïne Infusion on ad Libitum Food Intake and Satiety in Healthy Volunteers
Brief Title: Lidocaine and Food Intake
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: METC 163054
Record Dates: First submitted 2017-07-12; First posted 2017-07-24 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Hunger
MeSH Terms: interventions — Lidocaine; Water; Injections

STUDY DESIGN:
Intervention Model Description: Double blind randomized cross over trial
Who Masked: Participant, Investigator
Masking Description: Masking of participant and investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lidocaine (Active Comparator): LIdocaine dissolved in water for injections
  Interventions: Drug: Lidocaine
- Placebo (Placebo Comparator): Water for injections
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Lidocaine — Intragastric infusion of lidocain
  Arms: Lidocaine
Drug: Placebos — Intragastric infusion of water for injections
  Other Names: water for injections
  Arms: Placebo

SUMMARY:
World's population over 60 years old is increasing rapidly. It is expected that in 2050 elderly population will be 22% of the total population, representing around 2 billion people. This situation means a rising in the incidence of elderly-related diseases, and thereby the need for long-term care. Reduction in body fat and weight are a common problem among the institutionalized elderly. Some factors that contribute to the anorexia of aging are decreased perception of hunger and increased satiation. This represents an increased risk of developing cachexia even during minor illnesses. The potentially severe consequences of anorexia of aging a greater understanding of the underlying mechanism of these changes is highly important. Intraesophageal and intragastric infusion of 20mg/kg lidocaine results in an increase in food intake in Wistar rats. All infusions were done 30 minutes before the start of the meal intake (meal consisted of mealworms). It may be possible to decrease satiation, increase hunger, and hence food intake in elderly individuals through gastric infusion of the anesthetics lidocaine or benzocaine. In the future this study could potentially contribute to improve food intake in elderly vulnerable of losing body weight. Therefore, the current study aims to investigate the effect of intragastric administration of lidocaine on food intake, satiety/satiation and gastrointestinal complaints.

DETAILED DESCRIPTION:
Aim: To determine the effect of intragastric infusion of lidocaine on satiation, gastrointestinal complaints and food intake.

Hypothesis: We hypothesize that intragastric administration of lidocaine will result in a delay of postprandial satiation and hereby will result in an increase in food intake. Furthermore, lidocaine infusion will not result in an increase in any gastrointestinal complaints.

Primary objective: To investigate the effect of intragastric infusion of lidocaine on ad libitum food intake.

Secondary Objective(s):

1. To investigate the effect of intragastric infusion of lidocaine on satiety/satiation.
2. To study the effect of intragastric infusion of lidocaine on gastrointestinal complaints.

Design: Double blind randomized placebo-controlled cross-over trial in healthy male volunteers.

Study population: 35 healthy human male volunteers, 18 - 50 years old. Main study parameters/endpoints: Difference in ad libitum meal intake (as measured during ad libitum chili con carne meal).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Visual Analogue Scales (VAS) scores for satiety feelings (e.g., satiety, fullness, hunger, prospective feeding, desire to eat, desire to snack) and gastrointestinal symptoms (burning, bloating, belching, cramps, colics, warm sensation, sensation of abdominal fullness, nausea and pain) will be measured using VAS (0 to 100 mm) anchored at the low end with the most negative or lowest intensity feelings (e.g., extremely unpleasant, not at all), and with opposing terms at the high end (e.g., extremely pleasant, very high, extreme). Volunteers will be asked to indicate on a line which place on the scale best reflects their feeling at that moment. The scoring forms will be collected immediately so that they cannot be used as a reference for later scorings.

Catheter placement: the subjects will perceive mild discomfort during the placement of the catheter. Subjects can, at any time, come in contact with the investigator if any problems occur. All participants are healthy volunteers and we don't expect any health benefits or disadvantages.

ELIGIBILITY:
Inclusion Criteria:

* Based on medical history and previous examination, no gastrointestinal complaints can be defined.
* Age between 18 and 50 years. Several studies (see introduction) showed a difference in response to a meal between young and elderly people. Inclusion of elderly could interfere with the outcome of this study. Goal of this study is to investigate whether a difference in food intake can be found after intragastric infusion of a local anaesthetic. For this proof of concept study we therefore choose to include healthy male volunteers with a maximum age of 50 years.
* BMI between 20 and 25 kg/m2
* Weight stable over at least the last 6 months (≤5% weight change)

Exclusion Criteria:

* Females, because of their hormonal cycle and the possible influence of these hormones on eating behaviour.
* History of severe cardiovascular, respiratory, urogenital, gastrointestinal/hepatic, haematological/immunologic, HEENT (head, ears, eyes, nose, throat), dermatological/connective tissue, musculoskeletal, metabolic/nutritional, endocrine, neurological/psychiatric diseases, allergy, major surgery and/or laboratory assessments which might limit participation in or completion of the study protocol. The severity of the disease (major interference with the execution of the experiment or potential influence on the study outcomes) will be decided by the principal investigator.
* Use of amiodaron, because of the cardiotoxicity (in combination with lidocaine).
* Use of beta blockers, cimetidine and norepinephrine (synergetic effect on the action of Lidocaine).
* Other use of medication, which could interfere with the outcome of the study. This will be decided by the principal investigator.
* Administration of investigational drugs or participation in any scientific intervention study which may interfere with this study (to be decided by the principle investigator), in the 90 days prior to the study
* Major abdominal surgery interfering with gastrointestinal function (uncomplicated appendectomy, cholecystectomy and hysterectomy allowed, and other surgery upon judgement of the principle investigator)
* Dieting (medically prescribed, vegetarian, diabetic, macrobiological, biological dynamic)
* Excessive alcohol consumption (>20 alcoholic consumptions per week)
* Smoking
* Self-admitted HIV-positive state
* Any food allergy
* Not able to eat a chili con carne meal.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only males are eligible, because of the hormonal influence on food intake in females
Enrollment: 26 (Actual)
Dates: Start 2017-07-19 (Actual); Primary Completion 2018-06-26 (Actual); Study Completion 2018-06-26 (Actual)

PRIMARY OUTCOMES:
Difference in ad libitum meal intake after intragastric lidocain infusion compared to placebo | Difference between Test day 1 and Test day 2 (minimal wash out of 7 days)
  The difference in ad libitum food intake (kcal) after intragastric infusion of lidocaine and placebo and active within a subject.

SECONDARY OUTCOMES:
Difference in visual analogue scores for gastrointestinal complaints after intragastric lidocain infusion compared to placebo. | 15 minutes before the start of the infusion of placebo or lidocaine and after the start of the infusion every 15 minutes, until 90 minutes after start of infusion (8 times total).
  During a test day participants fill in 8 visual analogue scores (VAS) for gastrointestinal complaints (different time points). VAS scores will be recorded on a scale (0-100, 100mm) and will be measured.
Difference in visual analogue scores for satiation after intragastric lidocain infusion compared to placebo. | 15 minutes before the start of the infusion of placebo or lidocaine and after the start of the infusion every 15 minutes, until 90 minutes after start of infusion (8 times total).
  During a test day participants fill in 8 visual analogue scores (VAS) for satiation (different time points). VAS scores will be recorded on a scale (0-100, 100mm) and will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Ad Masclee, MD, PhD, Principal Investigator — Maastricht University Medical Center (MUMC+)
Locations (1):
- Maastricht University Medical Centre, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No